CLINICAL TRIAL: NCT00792727
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Four-Week Study to Assess the Efficacy and Safety of HKT-500 in Subjects With Pain Caused by Mild to Moderate Osteoarthritis of the Knee
Brief Title: HKT-500 in Adult Patients With Osteoarthritis (OA) Knee Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKT-500-US07
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: Pain; Knee; Arthritis; Knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen Patch (Experimental): Treatment with experimental drug
  Interventions: Drug: ketoprofen Patch
- Placebo Patch (Placebo Comparator): Treatment with placebo drug
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: ketoprofen Patch — 2 topical patches applied once daily for 28 days
  Other Names: Ketoprofen topical patch
  Arms: Ketoprofen Patch
Other: Placebo Patch — 2 topical placebo patches applied once daily for 28 days
  Other Names: Sham Treatment
  Arms: Placebo Patch

SUMMARY:
Ketoprofen in a topical patch formulation has been demonstrated to be effective for treating mild to moderate pain caused by various musculoskeletal disorders.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the short-term multiple dose efficacy and safety of HKT-500 in subjects with pain caused by mild to moderate osteoarthritis of the knee. The goal of the study is to gather additional information about the analgesic efficacy and safety of repeated, 24-hour applications of 2 HKT-500 patches per knee for a total of 28 days in subjects with pain caused by mild to moderate osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* man or woman ≥45 years of age.
* clinical diagnosis of unilateral or bilateral OA of the knee
* taking an NSAID or acetaminophen on a regular basis and has a history of knee pain amelioration with NSAID or acetaminophen use.
* mild to moderate OA of the knee at the screening visit
* subject exhibits an arthritis "flare" in the target knee within 7 days day of withdrawing from a NSAID or acetaminophen.
* subject understands that treatment will be administered on an inpatient basis.
* subject is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* subject is a woman of childbearing potential who has a positive urine pregnancy test, is lactating, or who is not surgically sterile
* subject has symptoms that are attributable to primary inflammatory diseases of the joint
* subject has unstable knees including a history of the knee catching or giving way or physical examination evidence of instability
* subject has arthropathies that occur in conjunction with systemic diseases
* subject has a chronic pain condition
* subject is grossly obese
* subject has a history of knee surgery within the past 12 months or arthroscopy within the past 6 months.
* subject has a history of osteotomies.
* subject is not willing to discontinue the use of NSAIDs, acetaminophen or other prohibited treatments
* subject used opioids for OA pain within 1 month

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change from the baseline of the WOMAC pain subscale score at Visit 6 (Day 14 ± 2 days) | 14 days ± 2 days

SECONDARY OUTCOMES:
WOMAC: Change from the baseline of the pain subscale score at Visit 5 (Day 7 ±1 day), Visit 7 (Day 21 ±3 days) and Visit 8 (Day 28 ±3 days) | 28 days (±3 days)
WOMAC: Change from the baseline of the subscale scores for stiffness and physical function at Visit 5, Visit 6, Visit 7 and Visit 8 | 28 days (±3 days)
WOMAC: Change from the baseline of the composite score at Visit 5, Visit 6, Visit 7 and Visit 8 | 28 days (±3 days)
Pain Intensity differences at rest, on motion and of overall assessment using a VAS scale at each follow-up assessments time point through Day 28. | 28 days
Subject's Global Assessment at Visit 6 and Visit 8 | 28 days (±3 days)
Investigator's Global Assessment at Visit 6 and Visit 8 | 28 days (±3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Kenichi Furuta, Study Director — Hisamitsu Pharmaceutical Co., Inc.
Locations (34):
- United States (34):
  - Hisamitsu Investigator Site, Birmingham, Alabama
  - Hisamitsu Investigator Site, Chandler, Arizona
  - Hisamitsu Investigator Site, Peoria, Arizona
  - Hisamitsu Investigator Site, San Diego, California
  - Hisamitsu Investigator Site, Colorado Springs, Colorado
  - Hisamitsu Investigator Site, Denver, Colorado
  - Hisamitsu Investigator Site, Daytona Beach, Florida
  - Hisamitsu Investigator Site, Delray Beach, Florida
  - Hisamitsu Investigator Site, Fort Myers, Florida
  - Hisamitsu Investigator Site, Pembroke Pines, Florida
  - Hisamitsu Investigator Site, Evansville, Indiana
  - Hisamitsu Investigator Site, Crestview Hills, Kentucky
  - Hisamitsu Investigator Site, Fall River, Massachusetts
  - Hisamitsu Investigator Site, Omaha, Nebraska
  - Hisamitsu Investigator Site, Las Vegas, Nevada
  - Hisamitsu Investigator Site, Reno, Nevada
  - Hisamitsu Investigator Site, Albuquerque, New Mexico
  - Hisamitsu Investigator Site, Greensboro, North Carolina
  - Hisamitsu Investigator Site, Bismarck, North Dakota
  - Hisamitsu Investigator Site, Cincinnati, Ohio
  - Hisamitsu Investigator Site, Columbus, Ohio
  - Hisamitsu Investigator Site, Mogadore, Ohio
  - Hisamitsu Investigator Site, Zanesville, Ohio
  - Hisamitsu Investigator Site, Oklahoma City, Oklahoma
  - Hisamitsu Investigator Site, Tulsa, Oklahoma
  - Hisamitsu Investigator Site, Warwick, Rhode Island
  - Hisamitsu Investigator Site, Anderson, South Carolina
  - Hisamitsu Investigator Site, Austin, Texas
  - Hisamitsu Investigator Site, San Antonio, Texas
  - Hisamitsu Investigator Site, Salt Lake City, Utah
  - Hisamitsu Investigator Site, Arlington, Virginia
  - Hisamitsu Investigator Site, Charlottesville, Virginia
  - Hisamitsu Investigator Site, Newport News, Virginia
  - Hisamitsu Investigator Site, Yakima, Washington